CLINICAL TRIAL: NCT04742751
Title: An Open-Label Pilot Intervention Trial to Prevent Diabetes in Prediabetic Adult Survivors of Childhood Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: St. Baldrick's Foundation (Other); Conquer Cancer Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PREDM; R21CA261713 (NIH)
Record Dates: First submitted 2021-01-06; First posted 2021-02-08 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: PreDiabetes; Adult Children
MeSH Terms: conditions — Prediabetic State | interventions — Metformin

STUDY DESIGN:
Masking Description: The schema was changed the to an adaptive trial design with a 12 week lifestyle run-in followed by a combined metformin+lifestyle intervention for 12 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Metformin is an antihyperglycemic agent which improves glucose tolerance in patients with type 2 diabetes mellitus, lowering both basal and postprandial plasma glucose. Metformin decreases hepatic glucose production, decreases intestinal absorption of glucose, and improves insulin sensitivity by increasing peripheral glucose uptake and utilization. With Metformin therapy, insulin secretion remains unchanged while fasting insulin levels and day-long plasma insulin response may decrease.
  Interventions: Drug: Metformin; Behavioral: Digital Intervention

INTERVENTIONS:
Drug: Metformin — To begin week 12 for participants who remain prediabetic after 12 week lifestyle run-in. Dosage and Route of Administration: 500 mg dose/ day to be taken orally, increased to 1000 mg dose/ day at week 14 through week 24. The dose should be taken immediately following the evening meal and at approximately the same time daily
  Other Names: D-Care DM2; Fortamet; Glucophage; Glucophage XR; Glumetza; Riomet; Metformin ER
Behavioral: Digital Intervention — Lifestyle Change Digital Intervention - This is a digital platform that will include a core curriculum focused on diet, exercise, and behavioral strategies for goal setting and self-monitoring to improve diet including a weight loss On Day 1, participants will begin their digital lifestyle intervention using their smart-phone application with their lifestyle coach and peer group.
  On day 14, participants will be contacted by phone (+/- 4 days, day 10 to 18) and adherence assessed using virtual pill counts via phone calls.
  At weeks 4, 8, 16 and 20 a phone-based pill count for adherence and adverse event symptom log will be completed and study medication dispensed.
  At week 12 (interim assessment) and 24 (study-end), the participant will return to St. Jude Children's Research Hospital (SJCRH) for an in-person assessment.
  The digital lifestyle change program will complete at week 24.
  Other Names: Lifestyle Change Digital Intervention

SUMMARY:
This is a first-in survivor, single-arm pilot study with the goal of establishing evidence of feasibility and safety of a combined pharmacologic (metformin) and lifestyle intervention (using an existing digital platform) to prevent diabetes in prediabetic adult survivors of childhood cancer.

Primary Objective

The primary aim of this proposal is to establish the feasibility and safety of a 24-week combined metformin + intensive lifestyle intervention among adult survivors with prediabetes (including a 12-week lifestyle alone run-in followed by 12-week combined intervention among survivors remaining prediabetic).

Primary endpoints of this trial will be adherence to 1) daily metformin administration and 2) completion of required core-curriculum of the lifestyle change intervention. Safety will be assessed using the Global Rating of Side Effects Burden

Secondary Objectives

The secondary aim is to assess preliminary evidence for efficacy of the combined metformin + intensive lifestyle intervention on glycemic control and insulin resistance. Glycemic control will be measured by fasting plasma glucose (FPG) and hemoglobin A1c (HbA1c) and insulin resistance measured by the homeostatic model assessment (HOMA-IR) and IGF- binding protein 1 (IGF-BP1; a measure of insulin sensitivity strongly correlated with euglycemic insulin clamp testing).

Exploratory Objectives

To assess preliminary evidence for efficacy of the combined metformin + intensive lifestyle intervention on weight, other anthropometric measures, blood pressure and lipid profile, physical activity (self-reported and as measured by accelerometer), frailty measures, and health-related quality of life (HRQOL). We will also assess diabetes development at future SJLIFE visits.

To assess measures of participation in the lifestyle change program as well as barriers to participation and medication adherence.

DETAILED DESCRIPTION:
Eligible subjects who meet inclusion criteria will be enrolled in a 12 week run-in period of the digital lifestyle intervention program. At the 12 week study visit, those who remain prediabetic will received metformin extended release daily, first at lower dose (500 mg/day) to minimize gastrointestinal side effects (diarrhea, nausea, flatulence, bloating), then escalated to a maximum dose of 1000 mg/day at week 14. The digitally delivered lifestyle change program will include a core curriculum focused on diet quality, food types, exercise and behavioral strategies for goal setting, and self- monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Investigators will recruit to enroll 55 survivors who are at least 18 but <45 years of age who participate in the St. Jude Lifetime Cohort Study (SJLIFE) and have been identified to have prediabetes defined as hemoglobin A1c (HbA1c)
* Participant in SJLIFE
* ≥18 and <45 years of age
* Prediabetic: fasting plasma glucose 105-125 mg/dL, hemoglobin A1c 5.7- 6.4% (either or both criteria may be present) According to institutional and NIH policy, the study will accession research participants regardless of sex and ethnic background. Institutional experience confirms broad representation in this regard.

Exclusion Criteria:

* Absence of treatment related diabetes risk. Survivors will be excluded if their cancer treatment required observation only, surgery alone not involving the abdomen or brain, radiation alone not involving the chest (pancreatic risk), abdomen or brain (e.g. retinoblastoma treated with enucleation alone, melanoma of an extremity treated with excision alone, neuroblastoma in an infant requiring observation only)
* Diabetes at baseline assessment: FPG ≥126 mg/dL, HbA1c ≥6.5% or previous diagnosis by a physician (except gestational diabetes that resolved post-partum)
* BMI <19 kg/m2
* Current metformin use (including for any period ≥30 days in the past 1yr)
* Known allergy to metformin
* Current use of other oral glucose lowering medications, non-insulin injectable diabetes medications or insulin (Appendix)
* Current participation in a lifestyle change program
* Chronic kidney disease ≥ stage IIIb (eGFR < 45 mL/min)
* Severe cardiovascular disease or recent intervention (NYHA class ≥2 or heart failure hospitalization in the past 6mo, Aortic stenosis, Heart block including LBBB or 3rd degree AV block, SBP >180 or DBP >105 mmHg, myocardial infarction or coronary revascularization in the past 1 month)
* Severe hepatic dysfunction: cirrhosis or AST/ALT >3 times upper limit of normal
* Pulmonary disease with dependence on oxygen or daily use of bronchodilators
* Weight loss >10% in the past 6 months
* Bariatric surgery in the past 2 years
* Pregnant, within 3 months post-partum, nursing, or planning to become pregnant
* Anemia: hematocrit <36% in males or <33% in females
* Ongoing alcohol or substance abuse using criteria from the AUDIT and DAST questionnaires (Appendix)
* Diagnosis of schizophrenia or other psychotic disorder
* Vision impairment limiting ability to interface with the digital program
* Unable to swallow medication
* Non-English speaking
* Cognitive impairment defined by IQ <80
* Current active cancer or undergoing treatment for active cancer

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Adherence for feasibility | 2 years
  Adherence to the intervention with 80% adherence to prescribed metformin and completion of 60% of the digitally-delivered core education curriculum through the lifestyle change platform.
Digitally-delivered core education curriculum through the lifestyle change platform | At end of Week 24
  Adherence will be monitored by completion logs of lessons
Safety and Adverse Events (Symptom Log including monitoring for AEs) | Week 4
  An Adverse Event Monitoring Log with Global Rating of Side Effects Burden
Safety and Adverse Events (Symptom Log including monitoring for AEs) | Week 8
  An Adverse Event Monitoring Log with Global Rating of Side Effects Burden
Safety and Adverse Events (Symptom Log including monitoring for AEs) | Week 12
  An Adverse Event Monitoring Log with Global Rating of Side Effects Burden
Safety and Adverse Events (Symptom Log including monitoring for AEs) | Week 14
  An Adverse Event Monitoring Log with Global Rating of Side Effects Burden
Safety and Adverse Events (Symptom Log including monitoring for AEs) | Week 16
  An Adverse Event Monitoring Log with Global Rating of Side Effects Burden
Safety and Adverse Events (Symptom Log including monitoring for AEs) | Week 20
  An Adverse Event Monitoring Log with Global Rating of Side Effects Burden
Safety and Adverse Events (Symptom Log including monitoring for AEs) | Week 24
  An Adverse Event Monitoring Log with Global Rating of Side Effects Burden
Drug adherence/Pill Counts | Week 2
  Adherence will be monitored by pill counts showing participant taking study drug, metformin ER, 80% of the time.
Drug adherence/Pill Counts | Week 4
  Adherence will be monitored by pill counts showing participant taking study drug, metformin ER, 80% of the time.
Drug adherence/Pill Counts | Week 8
  Adherence will be monitored by pill counts showing participant taking study drug, metformin ER, 80% of the time.
Drug adherence/Pill Counts | Week 12
  Adherence will be monitored by pill counts showing participant taking study drug, metformin ER, 80% of the time.
Drug adherence/Pill Counts | Week 16
  Adherence will be monitored by pill counts showing participant taking study drug, metformin ER, 80% of the time.
Drug adherence/Pill Counts | Week 20
  Adherence will be monitored by pill counts showing participant taking study drug, metformin ER, 80% of the time.
Drug adherence/Pill Counts | Week 24
  Adherence will be monitored by pill counts showing participant taking study drug, metformin ER, 80% of the time.

SECONDARY OUTCOMES:
Glycemic Control | Baseline to Week 24 (on campus labs at Baseline, Week 12 and 24)
  Glycemic Control will be measured by Change in Hemoglobin A1c
Glycemic Control | Baseline to Week 24 (on campus labs at Baseline, Week 12 and 24
  Glycemic Control will be measure by Change in Fasting Plasma Glucose

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Dixon, MD, MPH, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.tjude.org/protocols

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT04742751/Prot_SAP_000.pdf